CLINICAL TRIAL: NCT06294873
Title: Stool Sample Collection Study for Colorectal Cancer Test Research and Development
Brief Title: Stool Sample Collection Study
Status: Recruiting | Type: Observational
Sponsor: Innovis LLC (Industry)
Collaborators: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Innovis RD-2301
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: A screening device for the detection of colorectal and other aerodigestive tract cancers — DNA test to screen to detect colon cancer and precancerous lesions

SUMMARY:
The primary objective of this study is to obtain de-identified stool specimens from participants with colonoscopic biopsy-based histopathologic diagnosis of colorectal cancer (CRC) and/or a ≥1 cm colorectal polyp/adenoma/mass found during pre-enrollment colonoscopy that is of sufficient size to require surgical excision or complex colonoscopic polypectomy.

The samples will be used for the purpose of research and development of a new molecular diagnostic test for the detection of neoplasms of the aerodigestive tract.

DETAILED DESCRIPTION:
Participants providing written informed consent to participate in the study will be provided with a stool collection kit with multiple components. Participants will perform whole stool collection at home using a standardized whole stool collection device designed to fit over the toilet seat. The kit will also include a small, white-capped collection tube which participants will be instructed to use to collect a stool sample from the whole stool to allow for a fecal immunochemical test (FIT). In addition, the kit will contain an investigational device that includes a collection scoop and buffering solution. The investigational device will be used by participants to collect a stool sample from the whole stool. After the two (2) samples are collected from the whole stool, a buffering solution will then be poured over the remaining whole stool. The residual buffered whole stool, the sample in the small, white-capped collection tube (FIT) and the partial stool sample in the investigational collection device will be returned to the Sponsor in a self-shipping box, per the instructions provided to the participants.

All stool samples will be provided ≥7 days post-colonoscopy and prior to initiating bowel preparation for surgery, and/or neoadjuvant chemotherapy, radiation therapy, and/or follow-up therapeutic colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is a person ≥18 years of age.
2. Participant has a diagnosis of CRC, at any stage, or ≥1 cm colorectal polyp/adenoma/mass found during pre-enrollment colonoscopy that is of sufficient size to require surgical excision or complex colonoscopic polypectomy.
3. Participant understands the study procedures and can provide informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Participant has actively bleeding hemorrhoids.
2. Participant has active synchronous extra-colonic aerodigestive tract cancers (e.g., lung, esophagus, stomach, or pancreatic cancer).
3. Participant has a prior history of extra-colonic aerodigestive tract malignancy within the past 5 years.
4. Participant has a history of any inflammatory bowel disease.
5. Participant has familial adenomatous polyposis, hereditary non-polyposis colorectal cancer (Lynch) syndrome, or other hereditary cancer syndromes.
6. Participant has benign (non-pre-cancerous) polyps such as inflammatory polyps or hamartoma polyps.
7. Individual has a condition the Investigator believes would interfere with their ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women 18 years or greater with a diagnosis of CRC, at any stage, or ≥1 cm colorectal polyp/adenoma/mass found during pre-enrollment colonoscopy that is of sufficient size to require surgical excision or complex colonoscopic polypectomy.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Detection of colon cancer or precancer | 10 months
  To provide stool specimens to Exact Sciences to allow for additional research and development of a screening device for the detection of colorectal and other aerodigestive tract cancers.

CONTACTS AND LOCATIONS:
Overall Officials: Gregg S Britt, Study Director — Innovis LLC
Locations (3):
- United States (3):
  - Associated Gastroenterology Medical Group, Anaheim, California
  - Sarkis Clinical Trials, Ocala, Florida
  - Gastro One, Cordova, Tennessee

IPD SHARING:
Plan to Share IPD: No